CLINICAL TRIAL: NCT06466109
Title: Using Social Robots to Improve the Relationship and Alleviate Anxiety and Stress in Children With Rare Diseases and Their Parents: A Feasibility Study
Brief Title: Using Social Robots in Children With Rare Diseases and Their Parents: A Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-05-005B
Record Dates: First submitted 2024-05-24; First posted 2024-06-20 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Rare Diseases
Keywords: Robotics; Parent-Child Relations; Anxiety; Stress, Psychological; Rare Diseases
MeSH Terms: conditions — Rare Diseases; Anxiety Disorders; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: A single-group, pretest-posttest clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention group (Experimental): Patients and their parents will interact with the social robot PARO separately and together in each 30-minute course every two weeks for four courses.
  Interventions: Behavioral: social robot intervention

INTERVENTIONS:
Behavioral: social robot intervention — In the first and second courses, the patients and their parents freely interact with the social robot PARO for 30 minutes.
  In the third course, patients and their parents interact with PARO for 30 minutes using a worksheet that includes naming and recording characteristics of PARO.
  In the last course, patients and their parents interact with PARO for 30 minutes using a worksheet that freely recorded their observations about PARO and say goodbye to it.

SUMMARY:
The goals of this clinical trial are to (a) evaluate the feasibility and acceptability of a social robot intervention for providing family-based care for rare diseases families and (b) explore the effectiveness of the social robot intervention in improving the parent-child relationships and alleviating stress and anxiety for rare diseases patients and their parents. The main questions are:

* Is the social robot intervention suitable for and acceptable to rare disease patients and parents?
* Does the social robot intervention improve the parent-child relationship of rare disease patients and their parents?
* Does the social robot intervention alleviate the stress and anxiety of rare disease patients and their parents? Patients and their parents will interact with the social robot PARO separately and together in each 30-minute course every two weeks for four courses.

DETAILED DESCRIPTION:
Children with rare disease and their caregivers are distressed and stressed to deal with the disease and daily life, and their parent-child relationships are also challenging. Although social robots have been used to improve patients' and caregivers' well-being in clinical settings, there still needs to be family-centered, child-friendly, convenient, and feasible interventions for patients with rare diseases and their families. This study aims to evaluate the feasibility and acceptability of a social robot intervention for providing family-based care for rare disease families and explore the effectiveness of the social robot intervention in improving the parent-child relationships and alleviating stress and anxiety for rare disease patients and their parents. A single-group, pretest-posttest feasibility study will be conducted in two medical centers in Northern Taiwan. Of 21 dyads of 8- to 19-year-old children with rare diseases and their parents will be enrolled. The dyads will interact with the social robot PARO in each 30-minute course every two weeks for four courses. The retention rate will be calculated after the study, and the Friedman's test and Wilcoxon signed rank test will analyze the changes in the parent-child relationship, the anxiety, the perceived stress scales, and the heart rate variability. The content analysis will be used to analyze the interview data to delve into the child-parent-robot interaction and the effectiveness of the social robot intervention in the patients and the parents. This study is expected to provide a feasible and effective intervention to improve the psychological and social health of children with rare diseases and their caregivers and provide a reference for future randomized controlled trials of social robots in pediatric care.

ELIGIBILITY:
Inclusion Criteria:

[Patients]

* Aged 8 to 19 years.
* Diagnosed with a rare disease.
* Be Able to communicate in Chinese. [Parents]
* A father or a mother of a child with a rare disease.
* Be Able to communicate in Chinese.

Exclusion Criteria:

[Patients]

* Have a pacemaker.
* Have open wounds.
* Being infected with infectious diseases.
* Be unable to participate in social activities due to severe psychological disorder or cognitive dysfunction.

[Parents]

* Have a pacemaker.
* Have open wounds.
* Being infected with infectious diseases.
* Be unable to participate in social activities due to severe psychological disorder or cognitive dysfunction.

Ages: 8 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
retention rate | immediately after the intervention
  The retention rate is the average percentage of the patient-parent dyads who complete the 4-course intervention.
acceptability | immediately after the intervention
  The unified theory of acceptance and use of technology (UTAUT) scale will measure participants' acceptability of the social robot intervention. The chosen domains of this scale are perceived sociability (4 items), social presence (5 items), and perceived enjoyment (5 items) due to the importance of social robot interaction and sociability. Each item is assessed on a 5-point Likert scale, varying from 1 to 5; each domain's score is summed up individually; higher scores represent more agreement with this domain.
parent-child relationship | immediately after the intervention
  The elementary school student parent-child relationship scale will measure the patient's perceived parent-child relationship. The scale is composed of a 25-item questionnaire. Each item is assessed on a 5-point Likert scale, varying from 1 to 5, with total points ranging from 25 to 125, with higher scores representing better parent-child relationships.
  As for the parent's perceived parent-child relationship, the researcher modified part of the elementary school student parent-child relationship scale, and a psychological specialist validated the content. The score calculation is similar to the elementary school student parent-child relationship scale.
anxiety | immediately after the intervention
  The Chinese Version of the State Anxiety Scale for Children will measure the patient's anxiety. The scale is composed of a 20-item questionnaire. Each item is assessed on a 3-point Likert scale, varying from 1 to 3, with total points ranging from 20 to 60, with higher scores representing higher anxiety.
  The State-Trait Anxiety Inventory-State Anxiety will measure the parent's anxiety. The scale is composed of a 20-item questionnaire. Each item is assessed on a 4-point Likert scale, varying from 1 to 4, with total points ranging from 20 to 80, with higher scores representing higher anxiety.
stress | immediately after the intervention
  The heart rate variability and the Perceived Stress Scale will measure the patient's and the parent's stress. The researcher uses " Taiwan Scientific" Non-invasive Blood Pressure Meter to measure the heart rate variability, recording the low frequency power (LF), high frequency power (HF), and the ratio LF (ms2)/HF (ms2).
  The Perceived Stress Scale is composed of a 10-item questionnaire. Each item is assessed on a 5-point Likert scale, varying from 0 to 4, with total points ranging from 0 to 40, with higher scores representing higher perceived stress.

SECONDARY OUTCOMES:
child-parent-robot interaction | immediately after the intervention
  A self-designed questionnaire and an interview framework are used to explore the child-parent-robot interaction and the effectiveness of the social robot intervention in the patients and the parents individually. The 6-item questionnaire is assessed on a Visual Analogue Scale, ranging from 0 to 10. A higher score for each item represents being more engaged in the interaction with PARO, enjoying this intervention more, or being more willing to talk about the study with each other at home. The interview framework has six open-ended questions to delve into the patient's and the parent's experiences of the intervention.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - National Taiwan University Children's Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No